CLINICAL TRIAL: NCT06175117
Title: A Multicenter, Randomized, Double-blind, Parallel Controlled Clinical Study on the Efficacy and Safety of Compound E Jiao Jiang(cEJJ）in the Treatment of Postpartum Anemia
Brief Title: Clinical Study on the Treatment of Postpartum Anemia With Compound E Jiao Jiang(cEJJ）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongE E Jiao Coporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEEJ-CTP-20230724
Record Dates: First submitted 2023-11-27; First posted 2023-12-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- compound E Jiao Jiang(cEJJ) (Experimental): 20ml (1 bottle) at a time, 3 times a day, should be taken orally before morning, lunch and dinner.
  Interventions: Drug: compound E Jiao Jiang(cEJJ)
- compound E Jiao Jiang(cEJJ) placebo (Placebo Comparator): 20ml (1 bottle) at a time, 3 times a day, should be taken orally before morning, lunch and dinner.
  Interventions: Drug: compound E Jiao Jiang(cEJJ) placebo

INTERVENTIONS:
Drug: compound E Jiao Jiang(cEJJ) — compound E Jiao Jiang(cEJJ)：20ml (1 bottle) at a time, 3 times a day, should be taken orally before morning, lunch and dinner.
  Other Names: ferrous succinate tablet（1 tablet at a time, 2 times a day, should be taken in the morning, after dinner or during meals.）
  Arms: compound E Jiao Jiang(cEJJ)
Drug: compound E Jiao Jiang(cEJJ) placebo — compound E Jiao Jiang(cEJJ) placebo：20ml (1 bottle) at a time, 3 times a day, should be taken orally before morning, lunch and dinner.
  Other Names: ferrous succinate tablet（1 tablet at a time, 2 times a day, should be taken in the morning, after dinner or during meals.）
  Arms: compound E Jiao Jiang(cEJJ) placebo

SUMMARY:
The goal of this clinical trial] is to compare the effect of compound E Jiao Jiang(cEJJ）combined with iron decoction on postpartum anemia.The main questions it aims to answer are:

To evaluate the effectiveness of compound E Jiao Jiang(cEJJ） in the treatment of postpartum anemia.

To evaluate the safety of compound E Jiao Jiang(cEJJ） in the treatment of postpartum anemia.

To explore the effect of compound ejiao decoction on improving anxiety, depression, sleep and fatigue in postpartum anemia patients.

Participants will be randomly assigned (like flipping a coin) to either the trial group or the control group (with a 50% chance of being assigned to either group), where the trial group will receive the compound E Jiao Jiang(cEJJ） + ferrous succinate tablet, and the control group will receive the compound E Jiao Jiang(cEJJ）placebo + ferrous succinate tablet. The compound E Jiao Jiang(cEJJ）placebo is the same/similar to the compound E Jiao Jiang(cEJJ） in terms of appearance, smell and taste, but has no therapeutic effect.And participants need to return to the research center on time for relevant examinations according to the protocol requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild or moderate anemia (70g/L≤Hb < 110g/L) within 1 week postpartum and suitable for oral drug therapy;
2. Age 18-45 years old (including 18 and 45);
3. Those who do not use other iron agents and Chinese medicine/Chinese medicine preparations that have the effect of invigorating qi and nourishing blood during the study;
4. Sign the subject's informed consent voluntarily.

Exclusion Criteria:

1. Postpartum hemorrhage and blood transfusion treatment;
2. Those who received intramuscular/intravenous iron therapy or transfused blood products/human blood albumin and other plasma volume dilators within 3 months prior to screening;
3. Patients who have taken blood tonics within 1 week before screening, including other iron preparations and Chinese medicine or Chinese medicine preparations;
4. People with previous blood diseases such as sickle cell anemia, thalassemia, aplastic anemia, megaloblastic anemia;
5. Severe preeclampsia during pregnancy;
6. Abortion occurs in this pregnancy;
7. Patients with a serious digestive disease, cardiovascular disease, immune system disease, or serious mental disorder that the investigator believes may adversely affect the safety of the subject and/or the effectiveness of the investigational drug;
8. Severe hepatic and renal insufficiency (ALT >2×ULN, aspartate aminotransferase (AST)>2×ULN, Urea (Urea)/ urea nitrogen (BUN)>2×ULN, creatinine (Cr)>1×ULN);
9. Those who have a history of alcohol abuse, drug abuse or drug use before;
10. Allergic to the experimental drug or known ingredient;
11. Participants who had participated in other clinical trials within 3 months before screening;
12. Those who, according to the judgment of the investigator, consider it inappropriate to participate in this clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 360 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin（Hb） change value | 6 weeks
  Hb changes after 6 weeks of continuous medication

SECONDARY OUTCOMES:
The proportion of hemoglobin returned to normal | 6 weeks
  Hb returned to normal proportions after 6 weeks of continuous medication
The proportion of hemoglobin rising > 20g/L | 6 weeks
  The proportion of Hb increased >20g/L after 6 weeks of continuous administration
The proportion of hemoglobin rising > 10g/L | 6 weeks
  The proportion of Hb increased >10g/L after 6 weeks of continuous administration
serum iron change value | 6 weeks
  serum iron changes after 6 weeks of continuous medication
serum ferritin change value | 6 weeks
  serum ferritin changes after 6 weeks of continuous medication
Red Blood Cell（RBC） change value | 6 weeks
  RBC changes after 6 weeks of continuous medication
Hematocrit（HCT ）change value | 6 weeks
  HCT changes after 6 weeks of continuous medication
Traditional Chinese Medicine symptom score（a self-made scale for Qi-blood Deficiency Syndrome） change value | 6 weeks
  The TCM Qi and blood deficiency scale total score ranges from 0 to 54, and the higher the score, the more serious it is.

OTHER OUTCOMES:
Edinburgh Postnatal Depression（EPDS） change value | 6 weeks
  The EPDS total score ranges from 0 to 30, and the higher the score, the severe the depression.
Self-rating Anxiety Scale（SAS）change value | 6 weeks
  The SAS total score ranges from 0 to 80, and the higher the score, the greater the anxiety.
Pittsburgh sleep quality index（PSQI） change value | 6 weeks
  The PSQI total score ranges from 0 to 21, and the higher the score, the worse the sleep quality.
The Functional Assessment of Chronic Illness Therapy-Fatigue（FACIT-F） change value | 6 weeks
  The FACIT-F total score ranges from 0 to52, and the higher the score, the more fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical UniversityBeijing Maternal and Child Health Care Hospital, Beijing, China